CLINICAL TRIAL: NCT06299605
Title: Triple Versus Quadruple Therapy with Amoxicillin and Tetracycline for the Eradication of Helicobacter Pylori: a Multicenter Randomized Controlled Trial
Brief Title: Triple Versus Quadruple Therapy for the Eradication of Helicobacter Pylori
Acronym: SHARE2401
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Binzhou Maternal and Child Health Hospital (Unknown); Zibo Maternal and Child Health Hospital (Unknown); Zaozhuang Municipal Hospital (Other); Linyi Yizhou Hospital (Unknown); Feicheng Municipal People's Hospital (Unknown)
Responsible Party: Principal Investigator, Yanqing Li, Principal Investigator, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHARE2401
Record Dates: First submitted 2024-02-19; First posted 2024-03-08 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-03

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Tetracycline; Bismuth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 14-day quadruple regimen (Active Comparator): Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid + Bismuth 220mg bid for 14 days
  Interventions: Drug: Vonoprazan-Amoxicillin-Tetracycline-Bismuth quadruple regimen for 14 days
- 14-day triple regimen (Experimental): Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid for 14 days
  Interventions: Drug: Vonoprazan-Amoxicillin-Tetracycline triple regimen for 14 days
- 7-day triple regimen (Experimental): Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid for 7 days
  Interventions: Drug: Vonoprazan-Amoxicillin-Tetracycline triple regimen for 7 days

INTERVENTIONS:
Drug: Vonoprazan-Amoxicillin-Tetracycline-Bismuth quadruple regimen for 14 days — Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid + Bismuth 220mg bid for 14 days
  Other Names: Vonoprazan; Amoxicillin; Tetracycline; Bismuth; 14 days
  Arms: 14-day quadruple regimen
Drug: Vonoprazan-Amoxicillin-Tetracycline triple regimen for 14 days — Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid for 14 days
  Other Names: Vonoprazan; Amoxicillin; Tetracycline; 14 days
  Arms: 14-day triple regimen
Drug: Vonoprazan-Amoxicillin-Tetracycline triple regimen for 7 days — Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid for 7 days
  Other Names: Vonoprazan; Amoxicillin; Tetracycline; 7 days
  Arms: 7-day triple regimen

SUMMARY:
The study aimed to compare the efficacy and safety of 7-day and 14-day vonoprazan-amoxicillin-tetracycline triple therapy with 14-day vonoprazan-amoxicillin-tetracycline-bismuth quadruple therapy for the eradication of Helicobacter pylori. Subjects were randomized to receive the intervention and were reviewed by 13C-urea breath test after 6 weeks. The eradication rates, adverse reaction rates and patient adherence were calculated.

DETAILED DESCRIPTION:
H. pylori-positive patients without eradication history were recruited according to inclusion and exclusion criteria and randomized to the intervention:

14-day quadruple regimen: Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid + Bismuth 220mg bid for 14 days 14-day triple regimen: Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid 14 days 7-day triple regimen: Vonoprazan 20mg bid + Amoxicillin 1000mg bid + Tetracycline 500mg qid 7 days Subjects were asked to record adverse events and 6 weeks after treatment, 13C-urea breath test was tested for confirmation. The eradication rates, adverse reaction rates and patient adherence were calculated and analysed, and the results were analysed to provide more information for eradication regimens of H. pylori.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years old;
2. Patients with H.pylori infection (positive rapid urease test, 13C/14C-urea breath test);
3. Patients without previous treatment for H. pylori eradication.

Exclusion Criteria:

1. Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%;
2. Patients with active gastrointestinal bleeding;
3. Patients with a history of upper gastrointestinal surgery;
4. Patients allergic to treatment drugs;
5. Patients with medication history of bismuth, antibiotics within 4 weeks, or proton pump inhibitor within 2 weeks;
6. Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial;
7. Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse;
8. Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | Immediately after follow-up check
  13C-urea breath test was used to determine whether eradication was successful. Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in the three groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | Immediately after follow-up check
  A questionnaire on drug-related adverse reactions needs to be completed after treatment.
Patient compliance | Immediately after follow-up check
  A questionnaire on the number of missed and overdosed doses of medication needs to be completed after treatment. Good compliance was defined as taking 80%-120% of the pills.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Choi H, Leung K, Jiang F, Graham DY, Leung WK. Global prevalence of Helicobacter pylori infection between 1980 and 2022: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2023 Jun;8(6):553-564. doi: 10.1016/S2468-1253(23)00070-5. Epub 2023 Apr 20. PMID 37086739
- [Background] Crowe SE. Helicobacter pylori Infection. N Engl J Med. 2019 Mar 21;380(12):1158-1165. doi: 10.1056/NEJMcp1710945. No abstract available. PMID 30893536
- [Background] Malfertheiner P, Megraud F, Rokkas T, Gisbert JP, Liou JM, Schulz C, Gasbarrini A, Hunt RH, Leja M, O'Morain C, Rugge M, Suerbaum S, Tilg H, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study group. Management of Helicobacter pylori infection: the Maastricht VI/Florence consensus report. Gut. 2022 Aug 8:gutjnl-2022-327745. doi: 10.1136/gutjnl-2022-327745. Online ahead of print. PMID 35944925
- [Background] Lin K, Huang L, Wang Y, Li K, Ye Y, Yang S, Li A. Efficacy of genotypic susceptibility-guided tailored therapy for Helicobacter pylori infection: A systematic review and single arm meta-analysis. Helicobacter. 2023 Dec;28(6):e13015. doi: 10.1111/hel.13015. Epub 2023 Aug 27. PMID 37634236
- [Background] Savoldi A, Carrara E, Graham DY, Conti M, Tacconelli E. Prevalence of Antibiotic Resistance in Helicobacter pylori: A Systematic Review and Meta-analysis in World Health Organization Regions. Gastroenterology. 2018 Nov;155(5):1372-1382.e17. doi: 10.1053/j.gastro.2018.07.007. Epub 2018 Jul 7. PMID 29990487
- [Background] Jiang Z, Qian X, Wang Z, Dong Y, Pan Y, Zhang Z, Wang S. Antibiotic resistance of Helicobacter pylori isolated from patients in Nanjing, China: A cross-section study from 2018 to 2021. Front Cell Infect Microbiol. 2022 Sep 8;12:970630. doi: 10.3389/fcimb.2022.970630. eCollection 2022. PMID 36159644
- [Background] Chey WD, Megraud F, Laine L, Lopez LJ, Hunt BJ, Howden CW. Vonoprazan Triple and Dual Therapy for Helicobacter pylori Infection in the United States and Europe: Randomized Clinical Trial. Gastroenterology. 2022 Sep;163(3):608-619. doi: 10.1053/j.gastro.2022.05.055. Epub 2022 Jun 6. PMID 35679950
- [Background] Xie Y, Hu Y, Zhu Y, Wang H, Wang QZ, Li YQ, Wang JB, Zhang ZY, Zhang DK, Liu XW, Lu NH. Colloidal bismuth pectin-containing quadruple therapy as the first-line treatment of Helicobacter pylori infection: A multicenter, randomized, double-blind, non-inferiority clinical trial. Helicobacter. 2023 Jun;28(3):e12978. doi: 10.1111/hel.12978. Epub 2023 Mar 31. PMID 37002653